CLINICAL TRIAL: NCT04351906
Title: Low-flow Extracorporeal Carbon Dioxide Removal Using a Renal Replacement Therapy Platform for Correction of Hypercapnia in COVID-19-associated Acute Respiratory Distress Syndrome
Brief Title: Low-flow Extracorporeal Carbon Dioxide Removal in COVID-19-associated Acute Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ 63/20
Record Dates: First submitted 2020-04-09; First posted 2020-04-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: ARDS; Hypercapnic Respiratory Failure; AKI
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: ECCO2R
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECCO2R (Other): ECCO2R in patients with mild to moderate ARDS with/without AKI requiring dialysis.
  Interventions: Device: ECCO2R

INTERVENTIONS:
Device: ECCO2R — ECCO2R integrated into the multiFiltrate device

SUMMARY:
The study aims to investigate the efficacy of extracorporeal CO2 removal for correction of hypercapnia in coronavirus disease 19 (COVID-19)-associated acute respiratory distress syndrome

DETAILED DESCRIPTION:
The prevalence of acute respiratory distress syndrome (ARDS) caused by COVID-19 is approximately 8%. Lung-protective ventilation is the current standard of care for ARDS. It limits lung and distal organ impairment, but is associated with hypercapnia in approximately 14% of patients with mild to moderate ARDS and almost all patients with severe ARDS. In this setting, early implementing of an extracorporeal CO2 removal (ECCO2R) therapy may prevent further escalation of invasiveness of therapy (eg, need for extracorporeal membrane oxygenation (ECMO)). A number of low-flow ECCO2R devices are now available and some of those can be integrated into a renal replacement therapy (RRT) platform. This study aims to investigate the efficacy of an original ECCO2R system used in conjunction with a RRT platform in hypercapnic patients with COVID-19-associated mild-to-moderate ARDS with or without acute kidney injury (AKI) necessitating RRT.

ELIGIBILITY:
Inclusion Criteria:

* mild-to-moderate ARDS according to the Berlin definition
* lung-protective ventilation with positive end-expiratory pressure (PEEP) > 5 cm of water on mechanical ventilation expected to last > 24 h
* hypercapnia <80 mmHg
* bilateral opacities on chest imaging

Exclusion Criteria:

* age < 18 years
* pregnancy
* patients with decompensated heart failure or acute coronary syndrome
* respiratory acidosis with persistent partial pressure of blood carbon dioxide (PCO2) levels >80 mmHg
* acute brain injury
* severe liver insufficiency (Child-Pugh scores > 7) or fulminant hepatic failure
* decision to limit therapeutic interventions
* catheter access to femoral vein or jugular vein impossible
* pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-03 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Delta change in arterial partial pressure of carbon dioxide during ECCO2R treatment | Up to 72 hours
  Delta partial pressure of carbon dioxide change during ECCO2R treatment

SECONDARY OUTCOMES:
Change in vasopressor use during ECCO2R | Up to 72 hours
  Epinephrine and norepinephrine dose, mcg/kg/min
Assessment of changes in tidal volume during ECCO2R | Up to 72 hours
  Assessment of changes in tidal volume
Assessment of changes in pH during ECCO2R | Up to 72 hours
  Assessment of changes in pH
Assessment of changes in Positive End-Expiratory Pressure during ECCO2R | Up to 72 hours
  Assessment of changes in Positive End-Expiratory Pressure
Number of participants with adverse events directly related to ECCO2R | Up to 72 hours
  Adverse events directly related to ECCO2R are infection at the catheter site, hemorrhage at the cannulation site, air entry in the circuit.
Rate of technical adverse events related to ECCO2R | Up to 72 hours
  Adverse events directly related to ECCO2R are clotting of the circuit.
Delta change in venous partial pressure of carbon dioxide before and after ECCO2R membrane | Up to 72 hours
  Delta change in delta venous partial pressure of carbon dioxide before and after ECCO2R membrane

CONTACTS AND LOCATIONS:
Overall Officials: Werner Seeger, MD, Study Director — University Hospital Giessen and Marburg, Giessen
Locations (1):
- University Hospital Giessen and Marburg, Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schmidt M, Jaber S, Zogheib E, Godet T, Capellier G, Combes A. Feasibility and safety of low-flow extracorporeal CO2 removal managed with a renal replacement platform to enhance lung-protective ventilation of patients with mild-to-moderate ARDS. Crit Care. 2018 May 10;22(1):122. doi: 10.1186/s13054-018-2038-5. PMID 29743094
- [Derived] Husain-Syed F, Birk HW, Wilhelm J, Ronco C, Ranieri VM, Karle B, Kuhnert S, Tello K, Hecker M, Morty RE, Herold S, Kehl O, Walmrath HD, Seeger W, Vadasz I. Extracorporeal Carbon Dioxide Removal Using a Renal Replacement Therapy Platform to Enhance Lung-Protective Ventilation in Hypercapnic Patients With Coronavirus Disease 2019-Associated Acute Respiratory Distress Syndrome. Front Med (Lausanne). 2020 Nov 12;7:598379. doi: 10.3389/fmed.2020.598379. eCollection 2020. PMID 33304914